CLINICAL TRIAL: NCT01774656
Title: Remission From Stage D Heart Failure (RESTAGE-HF)
Brief Title: Remission From Stage D Heart Failure
Acronym: RESTAGE-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Principal Investigator, Emma Birks, M.D., Ph.D., University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTAGE-UL
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: heart-assist device
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HeartMate II plus Pharmacological Treat (Experimental): The HM II pump contains a single moving component, the rotor. The pump is implanted just below the left hemidiaphragm with the inflow attached to the apex of the left ventricle and the outflow graft anastomosed to the ascending aorta. Blood is pumped continuously throughout the cardiac cycle from the left ventricle to the aorta.
  The pharmacological treatment intended to enhance reverse remodeling includes 4 drugs initiated immediately after weaning of inotropic support once achieving adequate end-organ recovery and titrated (against symptoms, potassium, and renal function) to the following maximum doses: lisinopril 40 mg daily; carvedilol 25 mg 3 times daily; spironolactone 25 mg daily; digoxin 125g daily, and losartan 150 mg daily.
  Interventions: Drug: Pharmacological Treatment

INTERVENTIONS:
Drug: Pharmacological Treatment — The pharmacological treatment intended to enhance reverse remodeling includes 4 drugs initiated immediately after weaning of inotropic support once achieving adequate end-organ recovery and titrated (against symptoms, potassium, and renal function) to the following maximum doses: lisinopril 40 mg daily; carvedilol 25 mg 3 times daily; spironolactone 25 mg daily; digoxin 125g daily, and losartan 150 mg daily.

SUMMARY:
The purpose of this study is to determine the proportion of subjects who have sufficient improvement in ventricular function after undergoing a standardized Left Ventricular Assist Device (LVAD) plus pharmacologic recovery treatment and testing protocol to allow removal of the LVAD within 18 months.

DETAILED DESCRIPTION:
The encouraging results from the LVAD based recovery series suggest that the significant hemodynamic unloading provided by the Mechanical Circulatory Support (MCS) in conjunction with aggressive pharmacological treatment may induce a profound reverse structural remodeling and in turn result in a curative alternative to a specific patient population with severe heart failure. The active identification and characterization of the patients with a high potential for full cardiac function recovery is of paramount importance. The development of a standard and simplified recovery protocol would ultimately lead to a larger bridge to recovery patient population. The primary objective of this study is to determine the proportion of subjects who have sufficient improvement in ventricular function (remission from heart failure) after undergoing a standardized LVAD plus pharmacologic recovery treatment and testing protocol to allow removal of the LVAD within 18 months. The secondary objectives of this study are twofold, first to determine the durability of sustained remission from HF following LVAD explantation at 12 months and up to 3 years and second to determine the predictors of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age between 18 - 59 years, inclusive
2. Subject indicated for DT or BTT
3. Subject with severe clinical heart failure resistant to intensive medical therapy and requiring LVAD implantation
4. Subject with LVEF < 25% and cardiomegaly at the time of LVAD implantation as documented by radionuclide or contrast ventriculography or by echocardiography
5. Subject with non-ischemic etiology (confirmed by angiography either within 2 years of implantation or prior to explantation)
6. Subject have undergone HM II implantation within prior 4 weeks or planned for a HM II implant
7. Subject has a history of HF < 5 years.

Exclusion Criteria:

1. Subject has evidence of active acute myocarditis confirmed by histology
2. Subject has a history of previous CVA resulting in significant fixed motor deficit limiting ability to perform exercise testing
3. Subject has been implanted with a mechanical aortic and/or mitral valve(s)
4. Subject had an aortic valve closure
5. Subject diagnosed with a hypertrophic obstructive cardiomyopathy or sarcoidosis
6. Subject with LVEDD below normal confirmed by surface echocardiogram (restrictive cardiomyopathy)
7. Subject has irreversible multi-organ failure
8. Pregnant or lactating women or unwilling to utilize two reliable methods of birth control for women of childbearing age
9. Subject is diagnosed with a psychiatric disease, irreversible cognitive dysfunction or poor psychosocial issues that is likely to impair compliance with the study protocol
10. Subject with any condition, other than heart failure, that could limit survival to less than 2 years
11. Subject has a history of cardiac or other organ transplant
12. Subject is contraindicated to anticoagulation antiplatelet therapy
13. Subject requires acute or chronic renal replacement therapy (e.g. chronic dialysis) within 3 months prior to enrollment
14. Subject participating in any other clinical investigations involving another Mechanical Circulatory Support (MCS) device or heart failure related drug, or investigations which are likely to confound study results or affect study outcome.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who experience LVAD removal and subsequent freedom from mechanical circulatory support or heart transplantation | 12 months

SECONDARY OUTCOMES:
The proportion of evaluable subjects meeting explant criteria and subsequently explanted | 6 weeks, 3, 4, 5, 6, 9, 12-18 months
The time course of reverse remodeling on a left ventricular assist device | 6 weeks, 3, 4, 5, 6, 9, 12-18 months
The time course and sustainability of reverse remodeling following LVAD explantation | 12-18 months
Predictors of recovery and device removal | 6 weeks, 3, 4, 5, 6, 9, 12-18 months
Changes in maximal and sub maximal exercise capacity | 12-18 months
Changes in renal function and hepatic enzymes | 6 weeks, 3, 4, 5, 6, 9, 12-18 months
Changes in EF measured at 6000RPM. | 6 weeks, 4, 6, 9, 12-18 months
Changes in quality of life, as measured by the EuroQoL (EQ5D) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emma Birks, MD, Principal Investigator — University of Louisville
Locations (6):
- United States (6):
  - University of Louisville, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Birks EJ, Drakos SG, Patel SR, Lowes BD, Selzman CH, Starling RC, Trivedi J, Slaughter MS, Alturi P, Goldstein D, Maybaum S, Um JY, Margulies KB, Stehlik J, Cunningham C, Farrar DJ, Rame JE. Prospective Multicenter Study of Myocardial Recovery Using Left Ventricular Assist Devices (RESTAGE-HF [Remission from Stage D Heart Failure]): Medium-Term and Primary End Point Results. Circulation. 2020 Nov 24;142(21):2016-2028. doi: 10.1161/CIRCULATIONAHA.120.046415. Epub 2020 Oct 26. PMID 33100036